CLINICAL TRIAL: NCT00781300
Title: A Randomized Clinical Trial Comparing the Intraocular Pressure Changes With the Use of Loteprednol and Dexamethasone After Pterygium Surgery
Brief Title: Intraocular Pressure With Loteprednol and Dexamethasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Luciano Moreira Pinto, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 1104/03
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Intraocular pressure; Pterygium; Surgery; Steroids; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Pterygium; Glaucoma | interventions — Loteprednol Etabonate; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol (Active Comparator)
  Interventions: Drug: Loteprednol Etabonate 0.5%
- Dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone 0.1%

INTERVENTIONS:
Drug: Loteprednol Etabonate 0.5% — Patients in the Loteprednol Group received Loteprednol Etabonate 0.5% associated with Tobramycin 0.3% in separate eyedrops for four weeks: 6 times a day during the first postoperative week, 4 times a day during the second week, 3 times a day during the third week and twice-daily during the fourth week
  Other Names: Loteprol; Lotemax
  Arms: Loteprednol
Drug: Dexamethasone 0.1% — The patients in Dexamethasone Group received Dexamethasone 0.1% associated with Tobramycin 0.3% in a single eyedrop for four weeks: 6 times a day during the first postoperative week, 4 times a day during the second week, 3 times a day during the third week and twice-daily during the fourth week.
  Other Names: Tobradex
  Arms: Dexamethasone

SUMMARY:
The purpose of this study is to compare intraocular pressure (IOP) changes after pterygium surgery among patients using loteprednol and dexamethasone during the postoperative period.

DETAILED DESCRIPTION:
Surgical management of pterygium is known to initiate an inflammatory process with different levels of intensity. Corticosteroids are anti-inflammatory agents used to reduce the inflammatory process observed after surgical interventions including after pterygium surgery. However, use of topical corticosteroids can induce an elevation in intraocular pressure (IOP) due to a reduction in the facility of aqueous outflow.

Loteprednol etabonate (LE) was designed to maintain the anti-inflammatory efficiency of corticosteroids while lowering the risk of inducing IOP elevation. LE showed less effect on IOP than Prednisolone Acetate. This probably occurs due to lower levels of LE in the aqueous humor.

Some trials compare LE to other corticosteroids or placebo in treatments of the anterior uveitis, allergic conjunctivitis and cataract surgery. To our knowledge, there are no trials studying the effect of LE on IOP after pterygium surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: eighteen years old or more
* IOP: less than 22mmHg

Exclusion Criteria:

* History of previous ocular surgery
* Use of topical or systemic corticosteroids for up to a month before the surgery
* Extensive pterygia that disabled accurate IOP measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | Once a week for the first 4 weeks and 6 weeks after the procedure

SECONDARY OUTCOMES:
IOP difference between the operated eye and the fellow eye | Once a week for the first 4 weeks and then 6 weeks after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Luciano M Pinto, MD, Principal Investigator — Fedreal University of São Paulo
Locations (1):
- Department of Opthalmology, Federal University of São Paulo, São Paulo, São Paulo, Brazil